CLINICAL TRIAL: NCT06049914
Title: Combined Exercise and Nutrition Intervention for Possible Sarcopenia Among Community-dwelling Older Adults in Primary Care: A Randomized Controlled Trial
Brief Title: Combined Exercise and Nutrition Intervention for Possible Sarcopenia Among Older Adults in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Chang Won Won, Principal Investigator, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: KHMC-SARC-2023
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Elderly; Outpatient; Exercise; Intervention
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: 12-week combined exercise-nutrition intervention
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. Exercise interventions
     * Visiting the primary clinic twice a week and exercising at home once a week for a total of 6 weeks during the introductory and expanding period, and then visiting the primary clinic once a week and exercising at home twice a week for 6 weeks during the maintenance period
     * For exercise intervention, the researcher visits the primary clinic and conducts it face-to-face
     * Flexibility and strength Exercises: Up to 4 group exercises under the guidance of researchers, up to 40 minutes scheduled
  2. Nutritional interventions
     * Evaluate nutritional status through Mini Nutritional Assessment(MNA) survey at the time of Visit 1
     * Supplementary protein products are provided only for the malnourished group and at risk group with a MNA score of 23.5 or lower
     * Supplementary protein products: 'Mediwell', healthy five-grain flavor, liquid 150 ml, 150 kcal, 20g carbohydrates, 2g sugars, 8g protein, 5g fat
  Interventions: Behavioral: Experimental group
- Control group (No Intervention): * Control group: Providing only video and educational materials without intervention (12 weeks)
  * Videos and educational materials are provided to both the experimental group and the control group for home exercise.
  * Subjects write flexibility exercises, strength exercises, aerobic exercises, and meal diaries at home.

INTERVENTIONS:
Behavioral: Experimental group — 1. Exercise interventions
     * Measuring blood pressure and weight: before starting exercise
     * Flexibility exercises: 5-10 minutes of stretching
     * Strength exercises: Consists of 4 upper body exercises (Biceps Curl, Dips, Front raise, Chest press) and 5 lower body exercises (Leg lateral rotation, Leg extension, Hip abduction, Squat, Heel raise). The intensity of the band starts according to the subject's muscle strength.
     * Aerobic exercise: 5 times a week, home-based, 30 minutes or more each time
  2. Nutritional interventions
     * Well nourished: Overall diet check and correction
     * at risk: Correction of diet and intake of up to 2 packs of supplemental protein products per day
     * Malnourished: Correction of diet and intake of up to 3 packs of supplemental protein products per day
     * Nutrition counseling is provided at the beginning of the intervention and high-protein diet composition education is provided
     * Confirm compliance and provide feedback once every 2 weeks
  Arms: Experimental group

SUMMARY:
The purpose of this study is to assess the impact of a combined exercise-nutrition intervention in primary clinics on sarcopenia indices, physical function, and quality of life in community-dwelling older adults with possible sarcopenia.

DETAILED DESCRIPTION:
This study will investigate the effects of a 12-week combined exercise-nutrition intervention by comparing it with a control group receiving standard care (usual care) by assessing the sarcopenia indicators, functional recovery, and individual satisfaction. This is an interventional clinical study designed to recruit subjects, analyze data, identify problems, find improvement areas, and explore potential solutions.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 85 years of age
* Men and women with possible sarcopenia

  * If included in the possible sarcopenia criteria in the 2019 Asian Working Group for Sarcopenia(AWGS) criteria A Simple Questionnaire to Rapidly Diagnose Sarcopenia(The Korean SARC-F questionnaire) score is 4 or higher; or Calf circumference (Men's: <34 cm, Women's: <33 cm) + Decreased muscle strength (male: <28kg, female: <18kg) or Decreased physical function (if it takes more than 12 seconds from the 5-chair stand test)
  * [(1) and {(2) or (3)}]

Exclusion Criteria:

* Renal failure: Serum creatine exceeding 2.0 mg/dl
* Uncontrolled hypertension: systolic/diastolic blood pressure greater than 150/90 millimeter of mercury(mmHg)
* Uncontrolled diabetes: glycated hemoglobin (HbA1C) over 7.5%
* Subject who are receiving treatment (steroids, anticancer drugs, etc.) that can affect muscle mass
* Subjects with myocardial infarction or angina pectoris, stroke disease
* Malignant tumor: Subject who has a history of cancer within 5 years or is currently receiving treatment
* Subjects who have liver cirrhosis and uncontrolled hepatitis (Aspartate aminotransferase or Alanine aminotransferase is more than three times the upper limit of the reference range)
* Subjects who have chronic diseases such as musculoskeletal disorders that are impossible to exercise
* Subjects who are allergic to soybeans, coix, and brown rice

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
5-time chair stand test | Screening, 0st week of intervention, 6th week of intervention, 12th week of intervention
  a test of lower limb function that measures the fastest time taken to stand five times from a chair with arms folded.

SECONDARY OUTCOMES:
Grip strength | Screening, 0st week of intervention, 6th week of intervention, 12th week of intervention
  Measure maximum grip strength with a grip dynamometer
Falls | 0st week of intervention, 12th week of intervention, 24th week of intervention
  Falls Survey in Last 3 Months
EuroQol Visual Analogue Scale(EQ-VAS) | 0st week of intervention, 12th week of intervention
  a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Korean version of Instrumental Activities of Daily Living (K-IADL) | 0st week of intervention, 6th week of intervention, 12th week of intervention, 24th week of intervention
  Assess the skills and abilities needed to perform specific daily tasks related to an independent lifestyle in Korean version.
Korean version of Physical Activity Scale for the Elderly(K-PASE) | 0st week of intervention, 12th week of intervention
  Measures the level of self-reported physical activity in individuals aged 65 years or older and is comprised of items regarding occupational, household, and leisure activities during the previous 7-day period.
Mini Nutritional Assessment(MNA) | 0st week of intervention, 12th week of intervention
  Mini Nutritional Assessment is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition.
Korean version of Mini-mental State Examination(K-MMSE) | 0st week of intervention, 12th week of intervention
  a set of questions that commonly used to check for cognitive impairment (problems with thinking, communication, understanding and memory).
Korean version of Short Form of Geriatric Depression Scale(SGDS-K) | 0st week of intervention, 12th week of intervention, 24th week of intervention
  Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
The 12-item Health Survey(SF-12) | 0st week of intervention, 12th week of intervention
  Self-reported outcome measure assessing the impact of health on an individual's everyday life. It is used as a quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Won Won, MD, Principal Investigator — Kyunghee University Medical Center; Ja Euk Baek, Study Director — Dongdong Family Medicine Clinic; Seong Euk Kim, Study Director — Dongbu-hanil Surgery Clinic; Chung Hyeong Lee, Study Director — Seoulbom United Clinic; Mi Ji Kim, Study Director — Kyunghee University; Seon Yeong Kim, Study Director — Kyunghee University Medical Center; Jeong Ha Kim, Study Director — Chung-Ang University; Jeong Ha Park, Study Director — Kyunghee University Medical Center; Ga Yang Shim, Study Director — Kyunghee University Medical Center; Hye Suk Lee, Study Chair — Kyunghee University Medical Center; Dae Hyun Lee, Study Chair — Kyunghee University; Hee Eun Jung, Study Chair — Kyunghee University; Jae Young Jang, Study Chair — Kyunghee University; Na Hyun Lim, Study Chair — Kyunghee University; Hyun jin Cho, Study Chair — Kyunghee University; Min JIn Kim, Study Chair — Kyunghee University; Woohyuk Ji, Study Chair — Kyunghee University Medical Center
Locations (3):
- South Korea (3):
  - Dongdong Family Medicine Clinic, Dobong, Seoul
  - Dongbu-hanil Surgery Clinic, Dobong, Seoul
  - Seoulbom United Clinic, Dobong, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Research information will be provided to third parties (data processing organizations, academic societies, etc.) and used for secondary research. Individual participant data will be stored and used for 5 years after completion of the primary study. When used for secondary research, it will be used after deliberation by the institutional committee, and all information provided will be used only to create statistics for research purposes.
  The purpose and expected effect of third-party provision of research information and use of secondary research is to contribute to the promotion of national health.
  Personal information to be collected: Personal identification information (date of birth, name, gender, etc.), personal information (medical records necessary to determine the purpose of this study)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It will be distributed for storage/management/connection/provision for 5 years from the end of primary research by a data management agency determined by the Minister of Health and Welfare, and will be provided upon request by researchers for secondary research use only within that period.
Access Criteria: After deliberation by the institutional committee, it will be provided and utilized only for research that is judged to be of public interest through the Data Provision Deliberation Committee*.
  *Formation of a future data provision deliberation committee

REFERENCES:
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Arai H, Kritchevsky SB, Guralnik J, Bauer JM, Pahor M, Clark BC, Cesari M, Ruiz J, Sieber CC, Aubertin-Leheudre M, Waters DL, Visvanathan R, Landi F, Villareal DT, Fielding R, Won CW, Theou O, Martin FC, Dong B, Woo J, Flicker L, Ferrucci L, Merchant RA, Cao L, Cederholm T, Ribeiro SML, Rodriguez-Manas L, Anker SD, Lundy J, Gutierrez Robledo LM, Bautmans I, Aprahamian I, Schols JMGA, Izquierdo M, Vellas B. International Clinical Practice Guidelines for Sarcopenia (ICFSR): Screening, Diagnosis and Management. J Nutr Health Aging. 2018;22(10):1148-1161. doi: 10.1007/s12603-018-1139-9. PMID 30498820
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Jang HC. How to Diagnose Sarcopenia in Korean Older Adults? Ann Geriatr Med Res. 2018 Jun;22(2):73-79. doi: 10.4235/agmr.2018.22.2.73. Epub 2018 Jun 30. PMID 32743250
- [Background] Malafarina V, Uriz-Otano F, Malafarina C, Martinez JA, Zulet MA. Effectiveness of nutritional supplementation on sarcopenia and recovery in hip fracture patients. A multi-centre randomized trial. Maturitas. 2017 Jul;101:42-50. doi: 10.1016/j.maturitas.2017.04.010. Epub 2017 Apr 22. PMID 28539168
- [Background] Nipp RD, Fuchs G, El-Jawahri A, Mario J, Troschel FM, Greer JA, Gallagher ER, Jackson VA, Kambadakone A, Hong TS, Temel JS, Fintelmann FJ. Sarcopenia Is Associated with Quality of Life and Depression in Patients with Advanced Cancer. Oncologist. 2018 Jan;23(1):97-104. doi: 10.1634/theoncologist.2017-0255. Epub 2017 Sep 21. PMID 28935775
- [Background] Zhu LY, Chan R, Kwok T, Cheng KC, Ha A, Woo J. Effects of exercise and nutrition supplementation in community-dwelling older Chinese people with sarcopenia: a randomized controlled trial. Age Ageing. 2019 Mar 1;48(2):220-228. doi: 10.1093/ageing/afy179. PMID 30462162
- [Background] Yamada M, Kimura Y, Ishiyama D, Nishio N, Otobe Y, Tanaka T, Ohji S, Koyama S, Sato A, Suzuki M, Ogawa H, Ichikawa T, Ito D, Arai H. Synergistic effect of bodyweight resistance exercise and protein supplementation on skeletal muscle in sarcopenic or dynapenic older adults. Geriatr Gerontol Int. 2019 May;19(5):429-437. doi: 10.1111/ggi.13643. Epub 2019 Mar 13. PMID 30864254
- [Background] Chen HT, Wu HJ, Chen YJ, Ho SY, Chung YC. Effects of 8-week kettlebell training on body composition, muscle strength, pulmonary function, and chronic low-grade inflammation in elderly women with sarcopenia. Exp Gerontol. 2018 Oct 2;112:112-118. doi: 10.1016/j.exger.2018.09.015. Epub 2018 Sep 20. PMID 30243898
- [Background] Tsekoura M, Billis E, Tsepis E, Dimitriadis Z, Matzaroglou C, Tyllianakis M, Panagiotopoulos E, Gliatis J. The Effects of Group and Home-Based Exercise Programs in Elderly with Sarcopenia: A Randomized Controlled Trial. J Clin Med. 2018 Nov 26;7(12):480. doi: 10.3390/jcm7120480. PMID 30486262
- [Background] Lauque S, Arnaud-Battandier F, Mansourian R, Guigoz Y, Paintin M, Nourhashemi F, Vellas B. Protein-energy oral supplementation in malnourished nursing-home residents. A controlled trial. Age Ageing. 2000 Jan;29(1):51-6. doi: 10.1093/ageing/29.1.51. PMID 10690696
- [Background] Laddu D, Kim H, Phillips SA, Ma J. INERTIA: A pilot study of the impact of progressive resistance training on blood pressure control in older adults with sarcopenia. Contemp Clin Trials. 2021 Sep;108:106516. doi: 10.1016/j.cct.2021.106516. Epub 2021 Jul 24. PMID 34311098
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Derived] Ji W, Lee D, Kim M, Lim N, Lim JY, Baek JU, Kim S, Lee CH, Kim M, Won CW. Efficacy of a combined exercise and nutrition intervention study for outpatients with possible sarcopenia in community-based primary care clinics (ENdSarC): study protocol for a multicenter single-blinded randomized controlled trial. BMC Geriatr. 2024 Oct 23;24(1):861. doi: 10.1186/s12877-024-05434-y. PMID 39443873